CLINICAL TRIAL: NCT00142896
Title: Withdrawal Suppression Efficacy of Tramadol
Brief Title: Tramadol to Reduce Opioid Withdrawal Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Eric C. Strain/Principal Investigator, Johns Hopkins University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-18125-1; R01-18125-1; DPMC
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-08

CONDITIONS: Opioid-Related Disorders
Keywords: Opiate Addiction; Opiate Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Tramadol; Naloxone; Morphine

INTERVENTIONS:
Drug: Tramadol
Drug: Naloxone
Drug: Morphine

SUMMARY:
Individuals with opioid addiction often experience serious withdrawal symptoms that may make relapse unavoidable. Tramadol, a medication that is currently used to treat pain caused by chronic conditions such as cancer or joint pain, may also be effective at reducing opioid withdrawal symptoms. This study will evaluate the effectiveness of tramadol at reducing withdrawal symptoms in individuals addicted to opioid drugs.

DETAILED DESCRIPTION:
Opioid withdrawal symptoms are a major contributing factor for why opioid treatment programs often fail. Individuals with severe opioid withdrawal symptoms may experience shaking, muscle and bone pain, nausea, depression, anxiety, and drug craving. Tramadol is a medication that is currently used to treat moderate to severe pain in individuals with cancer, joint pain, or pain resulting from surgery. Because of its pharmacological profile, tramadol may also be useful in treating opioid withdrawal. Further research is needed to confirm the benefits of tramadol for opioid addicts. The purpose of this study is to evaluate the effectiveness of tramadol at reducing opioid withdrawal symptoms in opioid-dependent individuals.

This 6-week inpatient study will enroll opioid-dependent individuals. Participants will be required to reside at the research clinic for the entire study. All participants will receive morphine maintenance treatment on a daily basis. Twice a week participants will take part in experimental challenge sessions in which they will be randomly assigned to receive varying doses of tramadol, naloxone, morphine, or placebo. These sessions will assess the ability of tramadol to suppress opioid withdrawal symptoms. Participants will complete performance tasks to measure psychomotor and cognitive functioning. Heart rate and blood pressure will be monitored throughout the experimental sessions. A specialized camera will also be used to assess pupillary response of the eyes. Questionnaires and self-reports will be completed to assess medication effects and withdrawal symptoms. Following the end of the study, all participants will be offered outpatient drug abuse treatment.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV diagnostic criteria for opioid dependence
* Is in good physical health
* Qualifies for treatment with opioid agonist therapy (e.g., methadone)
* If female, must have a negative pregnancy test prior to study entry

Exclusion Criteria:

* Evidence of significant medical illness (e.g., insulin dependent diabetes mellitus)
* Evidence of significant psychiatric illness (e.g., schizophrenia)
* Currently seeking treatment for substance abuse
* Pregnant or breastfeeding

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2005-02; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Opioid withdrawal symptoms (measured by Visual Analog Scale during the experimental sessions)
Opioid agonist effects (measured by Visual Analog Scale during the experimental sessions)
Physiological effects (measured by pulse oximeter, blood pressure, heart rate, and pupillary camera during the experimental sessions)

CONTACTS AND LOCATIONS:
Overall Officials: Eric C. Strain, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (BPRU) Bayview Campus, Baltimore, Maryland, United States